CLINICAL TRIAL: NCT00953407
Title: Comparative Clinical Evaluation of Daily Disposable Lenses in Symptomatic Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-337-C-027
Record Dates: First submitted 2009-07-08; First posted 2009-08-06 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

ARMS (5):
- Nelfilcon A (Experimental): Nelfilcon A contact lens
  Interventions: Device: Nelfilcon A contact lens
- Narafilcon A (Active Comparator): Narafilcon A contact lens
  Interventions: Device: Narafilcon A contact lens
- Etafilcon A (Active Comparator): Etafilcon A contact lens
  Interventions: Device: Etafilcon A contact lens
- Omafilcon A (Active Comparator): Omafilcon A contact lens
  Interventions: Device: Omafilcon A contact lens
- Hilafilcon B (Active Comparator): Hilafilcon B contact lens
  Interventions: Device: Hilafilcon B contact lens

INTERVENTIONS:
Device: Nelfilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Nelfilcon A
Device: Narafilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Narafilcon A
Device: Etafilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Etafilcon A
Device: Omafilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Omafilcon A
Device: Hilafilcon B contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Hilafilcon B

SUMMARY:
The purpose of this trial is to evaluate the extent to which symptoms improve in symptomatic contact lens wearers when fit with one of 5 different daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Currently wear spherical, soft contact lenses replaced at intervals of 2 weeks or monthly.
* Habitually wear lenses for at least 8 hours per day, 4 days per week, for at least the past 6 months.
* Report 2 or more qualifying symptoms with current contact lenses with a frequency of "frequently" or "all the time"
* Able to achieve VA of at least 20/40 in each eye with habitual correction and with study lenses at dispense.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in any clinical trial.
* Any use of medications for which contact lens wear could be contraindicated as determined by the investigator.
* History of corneal refractive surgery.
* Cylinder correction greater than 1.00 D.
* Current monovision contact lens wearers.
* Other protocol inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled but not dispensed due to failing inclusion/exclusion criteria. These participants were included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Period: Overall Study
Arm/Group | Nelfilcon A | Narafilcon A | Etafilcon A | Omafilcon A | Hilafilcon B
Started | 26 | 25 | 26 | 25 | 24
Completed | 25 | 24 | 25 | 23 | 23
Not Completed | 1 | 1 | 1 | 2 | 1
Not completed — Failed inclusion criteria | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nelfilcon A: Nelfilcon A spherical contact lens worn on a daily wear, daily disposable basis
- Narafilcon A: Narafilcon A spherical contact lens worn on a daily wear, daily disposable basis
- Etafilcon A: Etafilcon A spherical contact lens worn on a daily wear, daily disposable basis
- Omafilcon A: Omafilcon A spherical contact lens worn on a daily wear, daily disposable basis
- Hilafilcon B: Hilafilcon B spherical contact lens worn on a daily wear, daily disposable basis
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A | Narafilcon A | Etafilcon A | Omafilcon A | Hilafilcon B | Total
Number analyzed (Participants) | 26 | 25 | 26 | 25 | 24 | 126
Age Continuous [Mean (Standard Deviation); unit: years] — This reporting group includes all enrolled and dispensed subjects.
  years | 29.5 (7.0) | 31.5 (11.9) | 29.9 (10.1) | 28.3 (7.7) | 30.5 (9.6) | 29.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — This reporting group includes all enrolled and dispensed subjects.
  Participants
    Female | 18 | 15 | 20 | 19 | 17 | 89
    Male | 8 | 10 | 6 | 6 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: Lens Awareness
Description: Lens awareness, as interpreted by the subject, was reported by the subject as a single, retrospective evaluation of 4 week's wear time. Frequency of lens awareness was measured on a 4-point scale, with 1 being never and 4 being all the time. Four-week ratings were compared to baseline ratings, and a negative difference (4-week minus baseline) represented an improvement.
Time Frame: 4 weeks of wear
Population: Per protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Number; unit: Participants
Arm/Group | Nelfilcon A | Narafilcon A | Etafilcon A | Omafilcon A | Hilafilcon B
Number analyzed (Participants) | 25 | 24 | 24 | 23 | 23
Participants | 16 (2.3) | 12 (2.8) | 11 (3.1) | 9 (2.5) | 13 (3.1)

ADVERSE EVENTS:
Time Frame: 8-1/2 weeks, duration of the study
Arm/Group | Nelfilcon A | Narafilcon A | Etafilcon A | Omafilcon A | Hilafilcon B
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/26 | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.